CLINICAL TRIAL: NCT00623077
Title: Dose Escalation of Total Marrow Irradiation Added to an Alkylator-Intense Conditioning Regimen for Patients With High Risk or Relapsed Solid Tumors
Brief Title: MT2004-30: Tomotherapy for Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Replaced by another study
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005LS023; UMN-MT2004-30 (Other: Blood and Marrow Transplantation Program); 0504M69306 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2008-02-22; First posted 2008-02-25 (Estimated); Last update posted 2017-12-05 (Actual); Status verified 2017-12

CONDITIONS: Brain and Central Nervous System Tumors; Kidney Cancer; Liver Cancer; Retinoblastoma; Sarcoma
Keywords: metastatic Ewing sarcoma/peripheral primitive neuroectodermal tumor; recurrent Ewing sarcoma/peripheral primitive neuroectodermal tumor; childhood hepatoblastoma; recurrent childhood liver cancer; stage IV childhood liver cancer; adult primary liver cancer; previously treated childhood rhabdomyosarcoma; recurrent childhood rhabdomyosarcoma; previously untreated childhood rhabdomyosarcoma; metastatic childhood soft tissue sarcoma; recurrent childhood soft tissue sarcoma; recurrent adult soft tissue sarcoma; stage IV adult soft tissue sarcoma; recurrent Wilms tumor and other childhood kidney tumors; stage IV Wilms tumor; stage V Wilms tumor; rhabdoid tumor of the kidney; stage IV renal cell cancer; childhood mixed glioma; recurrent childhood cerebellar astrocytoma; recurrent childhood cerebral astrocytoma; recurrent childhood ependymoma; recurrent childhood medulloblastoma; recurrent childhood pineoblastoma; recurrent childhood supratentorial primitive neuroectodermal tumor; recurrent childhood visual pathway glioma; untreated childhood brain stem glioma; untreated childhood cerebellar astrocytoma; childhood infratentorial ependymoma; childhood supratentorial ependymoma; childhood high-grade cerebellar astrocytoma; childhood high-grade cerebral astrocytoma; childhood low-grade cerebellar astrocytoma; childhood low-grade cerebral astrocytoma; newly diagnosed childhood ependymoma; childhood atypical teratoid/rhabdoid tumor; recurrent retinoblastoma; extraocular retinoblastoma; intraocular retinoblastoma; childhood renal cell carcinoma; clear cell renal cell carcinoma; recurrent renal cell cancer; recurrent childhood visual pathway and hypothalamic glioma; unspecified adult solid tumor, protocol specific; unspecified childhood solid tumor, protocol specific
MeSH Terms: conditions — Central Nervous System Neoplasms; Kidney Neoplasms; Liver Neoplasms; Retinoblastoma; Sarcoma; Neuroectodermal Tumors, Primitive, Peripheral; Hepatoblastoma; Carcinoma, Hepatocellular; Wilms Tumor; Carcinoma, Renal Cell; Astrocytoma; Familial ependymoma; Medulloblastoma; Optic Nerve Glioma; Rhabdoid Tumor | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; sargramostim; Busulfan; Etoposide; Ifosfamide; Melphalan; Thiotepa; Stem Cell Transplantation; Radiotherapy, Intensity-Modulated; Mesna

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Total Marrow Irradiation (MTI) with Tomotherapy (Experimental): TMI given prior to alkylator intensive conditioning regimen (Busulfan 9.6 mg/kg intravenously (IV) (>4 yrs of age) or 13.2 mg/kg IV (< 4 years of age), Melphalan 100 mg/m^2, Thiotepa 500 mg/m^2 for high risk solid tumor patients, Whole lung radiation 1500cGy in 10 fractions by Day 60, stem cell transplantation on day 0. Ifosfamide, etoposide, and mesna are given Days 0-4 followed by filgrastim for 3 doses. Cohorts of patients (n=3) will be treated with increasing doses of TMI (600, 1000, 1200 cGy) directed toward the bones.
  Interventions: Biological: filgrastim; Drug: busulfan; Drug: etoposide; Drug: ifosfamide; Drug: melphalan; Drug: thiotepa; Procedure: stem cell transplantation; Radiation: tomotherapy; Radiation: total marrow irradiation; Drug: Mesna; Radiation: Whole lung radiation

INTERVENTIONS:
Biological: filgrastim — Beginning 24 hours after chemotherapy end: 10 microgram/kg/day subcutaneously (SQ) or intravenously (IV) until absolute neutrophile count (ANC) > 1,000/mm^2.
  Starting that day, increase dose to 15 microgram/kg/day SQ or IV given as a single injection for 3 doses.
  Other Names: G-CSF; Sargramostim
Drug: busulfan — Part of pre-transplant conditioning chemotherapy: Administered as Busulfan 9.6 mg/kg IV (>4 yrs of age) or 13.2 mg/kg IV (< 4 years of age),every 6 hours on Days -8 through -6.
  Other Names: Busulfex; Myleran
Drug: etoposide — Part of Mobilization chemotherapy and Peripheral blood progenitor cell collections (day -100 to -30): Given as 100 mg/m^2/day intravenous (IV) over 1 hour for 5 days.
  Other Names: Eposin; VP-16
Drug: ifosfamide — Part of Mobilization chemotherapy and Peripheral blood progenitor cell collections (day -100 to -30): Given as 1.8 g/m^2/day intravenous (IV) over 1 hour on for 5 days.
  Other Names: Mitoxana; Ifex
Drug: melphalan — Part of pre-transplant conditioning chemotherapy: Administered as 100 mg/m^2 intravenous (IV) over 30 min on Days -5 through -4.
  Other Names: Alkeran
Drug: thiotepa — Part of pre-transplant conditioning chemotherapy: Administered as 500 mg/m^2 intravenously (IV) over 2 hrs on Days -3 through -2.
Procedure: stem cell transplantation — Regardless of whether the patient will be receiving peripheral cells or bone marrow, infusion will be intravenous on day 0, immediately after thawing.
  Other Names: HPC infusion
Radiation: tomotherapy — We plan to deliver the total marrow irradiation (TMI) to the upper half of the body using Tomotherapy TMI as explained in this protocol. However the lower part of the body will be treated with Anterior/Posterior linac based radiation treatment. Tomotherapy will then be delivered at a dose rate so as to keep the total treatment time to no more than 30 minutes. We anticipate that the dose rate will be around 400 cGy
  /minute (instantaneous dose rate).
Radiation: total marrow irradiation — TMI will be delivered to all bony sites as part of the conditioning. Additional "spot" therapy to PET positive lesions, primary disease (if not previously irradiated to maximum tolerated dose), and lungs will be performed on Day +60. Cohorts of 3 patients will be treated at a total dose of 600 cGy, 900 cGy or 1200 cGy on Days -11 through -9.
Drug: Mesna — Part of Mobilization chemotherapy and Peripheral blood progenitor cell collections (day -100 to -30): Given as 1.8 g/m^2/day divided in every 6 hrs dosing for 5 days.
  Other Names: Uromitexan®; Mesnex
Radiation: Whole lung radiation — At Day 60, patients with prior lung metastasis should receive whole lung irradiation (1500cGy in 10 fractions).

SUMMARY:
RATIONALE: A peripheral blood stem cell transplant or bone marrow transplant using stem cells from the patient may be able to replace immune cells that were destroyed by chemotherapy and image-guided intensity-modulated radiation therapy used to kill tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of bone marrow radiation therapy followed by an autologous stem cell transplant in treating patients with high-risk or relapsed solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the maximum tolerated dose of tomographic total marrow irradiation (TMI) when given prior to an alkylator-intensive conditioning regimen in patients with high-risk or relapsed solid tumors.

Secondary

* To determine the feasibility of performing positron emission tomography (PET) scans and spot radiation to PET-positive lesions after transplantation.
* To determine the change in bone mineral density and turnover in patients treated with an alkylator-intensive conditioning regimen and TMI.

OUTLINE:

* Mobilization chemotherapy and peripheral blood progenitor cell (PBPC) collection: Patients receive ifosfamide intravenously (IV) and etoposide IV on days -100 through -30.

Beginning 24 hours after completion of chemotherapy, patients receive filgrastim (G-CSF) subcutaneously (SC) or IV until blood counts recover. Patients then receive an increased dose of G-CSF SC or IV once daily for 3 consecutive days. Beginning on day -97, patients undergo up to 4 collections of PBPCs. Patients who do not yield an adequate number of cells undergo bone marrow harvest.

* Bone marrow harvest: Patients undergo bone marrow aspirate and biopsy 2 weeks after the last dose of G-CSF. If the aspirate or biopsy is morphologically free of tumor cells and demonstrates > 20% cellularity, then patients receive sargramostim (GM-CSF) daily for 5 days followed by bone marrow harvest.
* Total marrow irradiation (TMI) with tomotherapy: Patients undergo escalating doses of TMI* to all bony sites using helical tomotherapy image-guided intensity-modulated radiotherapy on days -11 to -9.

NOTE: *Patients with primary CNS tumors do not receive TMI but are eligible to receive chemotherapy and hematopoietic progenitor cell rescue in accordance with the protocol.

* Conditioning regimen: Patients receive busulfan IV over 2 hours four times daily on days -8 to -6, high-dose melphalan IV over 30 minutes on days -5 to -4, and thiotepa IV over 2 hours on days -3 to -2.
* Autologous CD34+ hematopoietic progenitor cell transplantation: Patients undergo reinfusion of autologous G-CSF-mobilized peripheral blood or bone marrow progenitor cells on day 0. Patients also receive G-CSF support beginning on day 0 and continuing until blood counts recover for 2 consecutive days.
* Post-transplantation radiotherapy: Patients may receive additional radiotherapy to areas of known metastatic disease, PET-positive lesions, primary disease (if not previously irradiated to maximum tolerated dose), and lungs beginning on day 60 post transplantation. Patients with prior lung metastasis may receive up to 10 fractions of whole-lung irradiation.

Patients may also receive additional radiotherapy to primary disease if maximum tolerated dose has not yet been reached.

Patients undergo bone mineral density studies at baseline and at days 60, 120, and 180 post transplantation. Patients also undergo blood sample collection periodically during study for pharmacokinetic analysis of busulfan.

Patients undergo PET scans at baseline and on day 60.

After completion of study therapy, patients are followed at days 180 and 365 and then periodically thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis Patients must have had histologic verification of malignancy at original diagnosis. Diseases included are:

  * Ewing's Family Tumors (ES/PNET/DSRCT): metastatic at the time of diagnosis and/or relapsed after therapy
  * Renal tumors: relapsed (all histology-Wilm's tumor) or at diagnosis (clear cell sarcoma and Rhabdoid tumor),
  * Hepatoblastoma: metastatic at the time of diagnosis and/or relapsed after therapy
  * Rhabdomyosarcoma: metastatic at the time of diagnosis and/or relapsed after therapy
  * Soft tissue sarcomas: chemotherapy responsive metastatic disease or chemotherapy responsive relapsed disease
  * Primary Malignant Brain Neoplasms at diagnosis and/or relapse
  * Retinoblastoma: disseminated at diagnosis and/or relapsed
  * Other High Risk Metastatic or Relapsed Solid Tumors: To be approved by two or more physicians on the study committee
* Disease Status: Patients must have either: 1) no evidence of disease or 2) stable, non-progressive disease (defined as non-progressive abnormalities on physical exam or computated tomography (CT) and/or magnetic resonance imaging [MRI]) within 4 weeks of study entry.
* Age: Patients must be 0-70 years of age at the time of study entry.
* Performance Level: Karnofsky > or = 50% for patients > 10 years of age and Lansky > or = 50% for patients < or = 10 years of age. Note: Neurologic deficits in patients with central nervous system (CNS) tumors must be stable for a minimum of 1 week prior to study entry.
* Organ Function:

  * Hematologic: prior to receiving total marrow irradiation (TMI) patients should have a hemoglobin of >10 gm/dl and a platelet count > 20,000/μl. Patients may receive transfusions as necessary.
  * Renal: glomerular flow rate (GFR) ≥ 50 ml/min/1.73m^2 or serum creatinine ≤ 2.5 x upper limit of normal (ULN) for age
  * Hepatic: aspartate aminotransferase/alanine aminotransferase (AST or ALT) ≤ 5 x ULN and bilirubin ≤ 5 x ULN
  * Cardiac: ejection fraction > 45% or no clinical evidence of heart failure
  * Pulmonary: oxygen saturation > 92% at rest (on room air)

Exclusion Criteria:

* Disease Status: patients with progressive, non-therapy responsive disease will not be eligible.
* Infection: patients who have active, uncontrolled infections or those who are HIV+.
* Pregnancy or Breast-Feeding: pregnant or breast-feeding women will not be entered on this study.
* Prior Radiation Therapy: patients must be eligible to receive TMI via tomographic radiation therapy (as determined by radiation oncology staff). If not eligible (due to extensive prior radiation or other circumstances), patients can be treated on study but will not receive radiation and will be analyzed on a separate arm.

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2005-08; Primary Completion 2012-07 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of tomotherapy up to 12 Gy | Day 42
  is a state-of-the- art means of delivering highly conformal radiation to tumors of targeted volume with high therapeutic gain. Tomotherapy offers unique advantages over total body irridiation and is expected to improve clinical outcome. The MTD is defined as the highest dose studied for which the incidence of dose limiting toxicity is less than 33%.

SECONDARY OUTCOMES:
Percent of patients who had PET scans and "spot radiation" to PET-positive lesions after transplantation | Day 60 Post Transplant
  PET-CT scan is done prior to and after transplant. Radiation is given before and after transplant.
Change in bone mineral density | Baseline, 6 and 12 Months Post Transplantation
  the change in bone density and turnover in patients exposed to alkylator intensive conditioning regimen followed by tomographic total marrow irradiation (TMI).
Rate of Treatment Related Mortality in Non-TMI Treated Patients | Day 100 Post Transplant
  Determined in patients who were not treated with total marrow irradiation; all deaths without previous relapse or progression are usually considered as related to transplantation.
Rate of Primary Neutrophil Engraftment | Day 42
  Neutrophil engraftment is defined as the first day of three consecutive days where the neutrophil count (absolute neutrophil count) is 500 cells/mm3 (0.5 x 109/L) or greater.
Overall Survival | From date of enrollment to date of death or censored at the date of last documented contact
  Determined in patients not receiving total marrow irradiation. The percentage of people in a study or treatment group who are alive for a certain period of time after they were diagnosed with or treated for a disease, such as cancer. Also called survival rate.
Disease-Free Survival | 1 Year
  In patients not receiving total marrow irradiation, the length of time after treatment ends that a patient survives without any signs or symptoms of that cancer or any other type of cancer. In a clinical trial, measuring the disease-free survival is one way to see how well a new treatment works.

CONTACTS AND LOCATIONS:
Overall Officials: Michael R. Verneris, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota, United States